CLINICAL TRIAL: NCT02756741
Title: Assessment of Cytokine Profile in an Open Labeled Randomized Controlled Trial of Standard Dose vs. Once a Day Intravenous Albumin in Patients With Spontaneous Bacterial Peritonitis
Brief Title: Comparison of Standard Dose Versus Once a Day Intravenous Albumin in Spontaneous Bacterial Peritonitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Subrat Kumar Acharya, Professor and Head, Department of Gastroenterology, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AIIMS sbp
Record Dates: First submitted 2016-04-24; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Cirrhosis
Keywords: Cirrhosis; hepatitis B virus; Alcohol; varices
MeSH Terms: conditions — Fibrosis; Hepatitis B; Varicose Veins | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- STANDARD DOSE (Active Comparator): Albumin 1.5gm/kg on day 1 and 1gm/kg on day 3
  Interventions: Drug: ALBUMIN
- LOW DOSE (Placebo Comparator): Albumin 20g/d for 5 days
  Interventions: Drug: ALBUMIN

INTERVENTIONS:
Drug: ALBUMIN — Albumin in two different doses

SUMMARY:
The standard recommended management of spontaneous bacterial peritonitis (SBP) includes a third-generation cephalosporin (cefotaxime or ceftriaxone) and high dose albumin (1.5g/kg on day 1 and 1g/kg on day 3). The major drawback of the current recommendations is the high price of albumin. In the current randomized control trial investigators compared the effect of standard recommended dose of albumin (1.5g/kg on day 1 and 1g/kg on day 3) vs. low dose (20g/d for 5 days) on the resolution of SBP and subsequent cytokine changes in ascitic fluid and blood.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of SBP
2. Age > 18 years
3. Consent to participate in the trial

Exclusion Criteria:

1. Secondary peritonitis
2. Malignancies including HCC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change in neutrophils/mm in ascitic fluid | 3 days
Change in IL-6, IL-1, TNF in ascitic fluid and serum between the two groups | 5 days

SECONDARY OUTCOMES:
Survival in days at the end of therapy | 5 days
Differences in frequency of sepsis, renal failure and other organ failures between the two groups | 5 days

IPD SHARING:
Plan to Share IPD: Yes